CLINICAL TRIAL: NCT01094223
Title: Mindfulness Based Relapse Prevention for Stimulant Users
Acronym: MBRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Suzette Glasner-Edwards, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBRP1R21DA029255-01
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Stimulant Dependence
Keywords: Stimulant; Addiction; Mindfulness; Treatment
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness (Experimental): Mindfulness Based Relapse Prevention (MBRP). Meditation based therapy group incorporating relapse prevention skills training.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention
- Health Education (Active Comparator): Health education, psychoeducation group focused on various topics pertaining to physical health
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention — Meditation based therapy group incorporating relapse prevention skills training
  Arms: Mindfulness
Behavioral: Health Education — Psychoeducation group focused on various topics pertaining to physical health
  Arms: Health Education

SUMMARY:
The broad, long-term objective of the current research is to improve treatment for stimulant use disorders by augmenting traditional relapse prevention therapy with innovative meditation-based strategies to promote affect regulation skills. Based on Mindfulness-Based Cognitive Therapy for depression (Segal, Teasdale, & Williams, 2002), Marlatt and colleagues recently developed a manualized intervention for the treatment of substance using populations: Mindfulness Based Relapse Prevention (MBRP). The specific aims of this research are 1) To conduct a pilot randomized clinical trial to assess the feasibility of recruiting and retaining individuals for a large scale study and to determine the effect size of MBRP relative to a health education (ED) control group in stimulant users receiving contingency management (CM).

DETAILED DESCRIPTION:
Both MBRP and ED participants will be assessed at baseline, treatment-end, and 1 month post-treatment. 2) To test the impact of MBRP compared to ED on negative affect, stimulant use, and health care outcomes. 3) To evaluate the differential effects of MBRP versus ED on HIV-risk behavior of participants, and 4) To examine potential mechanisms of action of MBRP, including reductions in stress reactivity and biological indicators of arousal such as blood pressure and heart rate. The investigators hypothesize that MBRP will be more efficacious than ED in reducing negative affect and stimulant use. Further, the investigators expect that MBRP will produce greater reductions in HIV-risk behaviors, stress reactivity, and arousal, and these changes will be associated with substance use outcomes. MBRP incorporates specific substance-focused cognitive therapy techniques with an additional emphasis on mindfulness skills. By providing coping skills to address affect regulation and stress reactivity, two important factors in stimulant relapse, MBRP may provide a promising augmenting strategy for the treatment of stimulant users.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 59
2. DSM-IV diagnosis of Stimulant Dependence
3. Able to provide informed consent
4. Willing and able to participate in study procedures

Exclusion Criteria:

1. Presence of life threatening or unstable medical illness, such as acute pulmonary, cardiovascular, or musculoskeletal disease, that would require treatment or make study participation difficult
2. Lack of proficiency in English
3. Currently homeless (unless residing in a recovery home for which contact information can be provided)
4. Dependence on an illicit substance for which medical detoxification is imminently needed.
5. Presence of clinically significant psychiatric symptoms as assessed by MINI, such as psychosis or acute mania, that would require ongoing treatment or make study compliance difficult.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | baseline (week 0), weekly during treatment (weeks 1-12), and at follow-up (week 24)
  The Beck Depression Inventory (BDI), a well validated self-report measure (Beck, 1967) will be administered at baseline, weekly during treatment, and at follow-up. Both the absolute total scores and change scores will be used for analyses.

SECONDARY OUTCOMES:
HIV Risk behaviors | baseline (week 0), treatment-end (week 12), and follow up (week 24)
  The HIV Risk Assessment Battery (Navaline et al., 1994) will be administered at baseline, treatment-end, and FU to assess the impact of the interventions on changes in HIV/AIDS-related risk behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Glasner, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States